CLINICAL TRIAL: NCT02898064
Title: Back Pain Prevention in Multiple Myeloma Using an External Spinal Brace - a Feasibility Study
Brief Title: Back Pain Prevention in Multiple Myeloma Using an External Spinal Brace
Acronym: MAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1017
Record Dates: First submitted 2016-06-29; First posted 2016-09-13 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care + brace (Other): Spinal brace (thoracolumbosacral orthosis or cervico-thoraco-lumbar orthosis) to be fitted to the participant in addition to receiving standard of care treatment which can include radiotherapy, chemotherapy or surgery including vertebral augmentation and also medication including bisphosphonates
  Interventions: Device: thoracolumbosacral orthosis or cervicothoracolumbar orthosis; Other: Standard care
- Standard care (Other): Participant will receive standard of care treatment which can include radiotherapy, chemotherapy or surgery including vertebral augmentation and also medication including bisphosphonates
  Interventions: Other: Standard care

INTERVENTIONS:
Device: thoracolumbosacral orthosis or cervicothoracolumbar orthosis — An "off the shelf spinal brace" which will be applied to the patients trunk. They will have straps and harnesses which the patient can fasten and remove if needed. The brace will need to be worn by the intervention group all the time for 3 months except when lying in bed. In the presence of lower thoracic (T8 downwards), thoraco-lumbar and lumbar (L1- L3) fractures, a thoracolumbosacral orthosis will be applied. For upper thoracic fractures (T1-T7) a cervico-thoracic or cervico-thoraco-lumbar orthosis will be used.
  Other Names: spinal brace
  Arms: Standard care + brace
Other: Standard care — Standard surgery, radiotherapy, chemotherapy, drug therapy as applicable and decided by the participants consultant as part of standard care

SUMMARY:
Consenting patients with multiple myeloma (MM) will be randomly allocated to receive either standard medical treatment (chemotherapy, radiotherapy, pain-killing medication) alone or standard medical treatment plus a brace. Patients will be regularly evaluated in research clinics; the results data will inform the design of a full trial. Information will be collected to inform a list of requirements a centre needs to have in place to run an RCT of these interventions.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a neoplasia of plasma cells mostly within the bone marrow, commonly leading to multiple vertebral collapses. This causes spinal deformity, leading to incapacitating back pain and reduced quality of life. In spite of advances in medical therapy, some patients are left with disabling back pain, sometimes requiring surgical intervention. University Hospitals of North Midlands NHS Trust have observed on an audit of our own practice that application of an external spinal brace as early in the disease process as is possible appears to maintain the overall alignment of the spine, thus minimising risk of spinal deformity and consequent back pain.

The ultimate aim is to undertake an RCT to determine whether the use of an external spinal brace can reduce back pain and spine-related disability in patients suffering from back pain due to multiple myeloma, in comparison to conventional management without a brace.

However, prior to this, a feasibility study is required. The feasibility study is needed to see if the trial processes (providing patient information, consent process, conducting the baseline investigations and outcome measures) can be accommodated without causing too much delay to the application of the brace.

Suitable patients will be consented by the research team and randomised to receive a brace or no brace in addition to their routine Myeloma treatment. After baseline data collection and questionnaires, the participant would be followed up for data collection at 6 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with MM
* Myeloma infiltration in the spine confirmed by radiological evidence
* MM-related back pain
* Can attend for the whole follow up period

Exclusion Criteria:

* Presenting with cord compression and neurological deficit requiring urgent decompression and intervention
* Chronic pain syndrome
* Language barrier that cannot be overcome using translation services
* Unwilling or unable to give informed consent
* Painful VCFs at the lumbosacral junction, L4 to Sacrum, where application of brace is not possible.

Not suitable for treatment with a brace e.g. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Time from diagnosis to brace fitting for patients randomised to the intervention group | Assessed at 3 months
Number of patients in the intervention arm who request additional support from the orthotic team and time they had to wait for support. | assessed at the end of study at 21 months
The number of orthotists in each hospital | 21 months
Are appropriate braces fitted | 6 weeks
  The locations and levels of VCFs and back pain in patients and the type of brace fitted will be recorded to determine whether appropriate braces are fitted.
Number of appointments issued by orthotists | 21 months
Frequency of appointments issued by orthotists | 21 months

SECONDARY OUTCOMES:
The number of new MM cases at each centre | 1 year
The number of eligible patients who give consent to enter the study | 21 months
The number of patients that drop-out during follow-up and their reasons | 21 months
The number of missing cases for a subsequent RCTs co-primary outcomes of pain and disability | 21 months
Pain measured by VAS | 6 weeks and 3 months
Descriptive statistics and qualitative analysis of the 3-month follow up patient questionnaire | 3 months
  The questionnaire consists principally of ordinal rating scales, which will be analysed descriptively in terms of frequencies, medians and interquartile ranges. Qualitative data from the supplementary open-ended questions will be analysed by means of framework analysis.
Qualitative assessment of semi structured interviews in a sub-set of participants, EQ-5D-5L | 21 months
The number of patients who receive non-study-related interventions during the 3 month follow-up period | 3 months
Disability measured by ODI | 6 weeks and 3 months
Number of patients eligible for the study during 1 recruitment year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Konduru, Study Director — University Hospitals of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised patient data would be published